CLINICAL TRIAL: NCT07185867
Title: Prevention of ANxiety and Depression Over Risk Assessment: a Randomized Controlled Trial (the PANDORA-Predict-Plus-Prevent Study)
Brief Title: Prevention of ANxiety and Depression Over Risk Assessment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Mediterranean Institute for the Advance of Biotechnology and Health Research (Other)
Collaborators: European Regional Development Fund (Other); Research Network on Chronicity, Primary Care, and Health Promotion (Unknown); Carlos III Health Institute (Other Government); IBIMA Plataforma BIONAD (Unknown); Andalusian Regional Ministry of Health (Other Government)
Responsible Party: Principal Investigator, Juan Ángel Bellón, PhD, Medicine, Andalusian Health Service
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PI21/01695
Record Dates: First submitted 2025-09-15; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Depression; Anxiety; Prevention; m-Health
Keywords: Depression; Anxiety; Prevention; Randomized Controlled Trial; m-Health; App; Predictive risk algorithms
MeSH Terms: conditions — Depression; Anxiety Disorders; Alzheimer Disease | interventions — Drug Interactions

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Pandora-1 app intervention (Experimental): In this arm, participants will use an internet-based, self-guided and personalized intervention to prevent depression and anxiety, which also includes risk predictive algorithms, personalized prevention plans, decision support systems, monitoring and feedback.
  Interventions: Behavioral: Pandora-1 app with high levels of personalization, interaction, monitoring and feedback
- Pandora-2 app intervention (Experimental): In this arm, participants will use an internet-based and self-guided intervention that includes psychoeducational brochures for the prevention of anxiety and depression that can be used when they want.
  Interventions: Other: Pandora-2 app with low levels of personalization, interaction, monitoring and feedback
- Control Condition (usual care) (No Intervention): Participants in this arm, as is also the case with participants in the Pandora-1 and -2 arms, will continue to receive usual care from their health providers and will fill out the same questionnaires and reminders. However, they will not receive information about their responses or suggestions related to them, except those included in the security protocol on suicide risk and potential clinical diagnosis of anxiety disorders or depression.

INTERVENTIONS:
Behavioral: Pandora-1 app with high levels of personalization, interaction, monitoring and feedback — Pandora-1 is a behavioral, self-guided and transdiagnostic intervention delivered via an app. It includes predictive risk algorithms, decision support systems (DSS), monitoring and feedback to implement personalized prevention plans (PPP) for anxiety and depression. The intervention has a biopsychosocial approach and offers 4 interactive modules: move more, sleep better, improve relationships and emotional well-being. Participants will receive personalized feedback at baseline, 1, 6 and 12 months, including their levels of depressive and anxiety symptoms over the past two weeks, their predicted risk of developing these disorders in the next year, and related modifiable risk factors (e.g. sedentary lifestyle, insomnia, low social support, poor mental quality of life). Based on this, the app offers suggestions (via DSS) and guides users to relevant content (PPP). Participants follow recommendations of choice, the app tracks these actions and provides feedback at baseline, 1 and 6 months.
  Arms: Pandora-1 app intervention
Other: Pandora-2 app with low levels of personalization, interaction, monitoring and feedback — Pandora-2 is a psychoeducational self-guided and transdiagnostic intervention delivered via an app. This intervention also has a biopsychosocial orientation and includes a set of psychoeducational brochures for the prevention of anxiety and depression that can be used at any time. These read-only brochures will have contents on the same 4 intervention modules (move more, sleep better, improve relationships and emotional well-being). At baseline, 1 and 6, 12 months participants will also receive basic information about their level of depressive and anxiety symptoms over the past two weeks, their risk probability of depressive and anxiety episodes next year and some of their modifiable risk factors associated with such risk (e.g. sedentary lifestyle, insomnia, low social support and poor mental quality of life). However, in Pandora-2 intervention participants will have lower levels of interactive intervention components as suggestions from the DSS about PPP, monitoring and feedback.
  Arms: Pandora-2 app intervention

SUMMARY:
The general goal is to design, develop and evaluate a personalized, self-guided and trans-diagnostic internet-based intervention to prevent anxiety and depression, based on predictive risk algorithms and decision support systems (DSS), in Spanish and Chilean adult population.

Methods: We will conduct a three-arm parallel randomized controlled trial with one year of follow-up. A total of 2,595 depression- or/and anxiety-free participants (865 per group), aged 18-65, will be recruited and randomly assigned to one of two intervention groups or to the usual-care group (in a 1:1:1 ratio). Both interventions, Pandora-1 and Pandora-2, will be implemented via a smartphone application, the Pandora App. Pandora-1 is a self-guided and transdiagnostic intervention that includes 4 interactive intervention modules (move more, sleep better, improve relationships and emotional well-being), as well as predictive risk algorithms, decision support systems, and monitoring and feedback to implement personalized plans for the prevention of anxiety and depression. Pandora-2 is a psycho-educative intervention with predictive risk algorithms, minimally interactive and without personalization. The primary outcome is the combined rate of the onset of anxiety or depression (DSM-V diagnoses as measured by the CIDI interview) at 6 and 12 months. The secondary outcomes are the reduction of depressive (PHQ-9) and anxious (GAD-7) symptoms, risk of depression and anxiety (predictD and predictA risk algorithms), and the improvement of mental & physical quality of life (SF-12), as well as acceptation and satisfaction with Pandora apps (u-MARS) and adverse effects (ad hoc questionnaire), which will be assessed at 1, 6 and 12 months. As mediators will be measured social support (Duke-UNC-2 items), physical activity (BPAQ-2), sleep (AIS-5), and repetitive negative thinking (PTQ-9) evaluated at 1, 6 and 12 months. We will use ActiGraph-GT3X accelerometers to assess physical activity and sleep at 1 and 6 months, in a subsample of 404 sedentary study participants.

DETAILED DESCRIPTION:
The specific goals are: 1) to adapt the epD-Work App (an App developed to prevent depression in the workplace with predictive risk algorithms, decision support system, monitoring and feedback, repositories, communication systems and intervention modules) in a new App, the Pandora App, for the personalized anxiety and depression prevention in Spanish and Chilean adult population; 2) to evaluate the usability and adherence of the participants to the Pandora interventions; 3) to evaluate the acceptability and satisfaction of the participants regarding the Pandora interventions; 4) to evaluate the effectiveness of the Pandora interventions to reduce the onset of episodes of major depression and anxiety disorders; 5) to evaluate the effectiveness of the Pandora interventions in reducing depressive and anxious symptoms and the probability of developing depression and anxiety in the next 12 months (predict-D and predict-A risk algorithm); 6) to evaluate the effectiveness of the Pandora interventions to improve physical and mental quality of life; 7) to perform a causal analysis on the anxiety and depression preventive effect of the Pandora intervention taking into account several mediators and moderators; and 8) to evaluate the appearance of undesirable effects associated with the use of the Pandora interventions.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent acceptance
* Having a valid telephone number
* Ownership of an Apple-Android-operating smartphone with an internet connection
* 18-65 years old
* Habitually reside (> 6 months/year) in Spain or Chile

Exclusion Criteria:

* Difficulty reading and/or understanding Spanish
* Suffer from disabling neurological conditions (dementia, blindness, etc.) that makes it difficult to use smartphone, terminal illness with a life expectancy < 12 months, a history of severe mental disorders confirmed by a healthcare professional (schizophrenia or psychosis, bipolar, anoxeria, bulimia or personality disorders), having alcohol or substance use disorder within the past year
* Currently receiving face to face or via internet psychological treatment (currently taking antidepressants or anxiolytics is not an exclusion criterion, but their use will be taken into account throughout the follow-up)
* Presence of clinically relevant anxiouys (GAD-7 score ≥ 10 points) or depressive symptoms (PHQ-9 score ≥ 10 points).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2595 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2028-03-07 (Estimated); Study Completion 2028-03-07 (Estimated)

PRIMARY OUTCOMES:
Combined onset of depression-anxiety event | 6 and 12 months follow-up
  The primary outcome of this study will be a combined onset of depression-anxiety event (yes/no) as endpoint, which will include the following DSM-V diagnoses: major depressive disorder, generalized anxiety disorder, panic disorder, agoraphobia and social phobia as measured by standardized psychiatric interview (CIDI: Composite International Diagnostic Interview).

SECONDARY OUTCOMES:
Depressive symptoms (PHQ-9) | Base line, 1, 6 and 12 months follow-up
  Depressive symptoms will be measured by the PHQ-9, which is a reliable and valid 9-item measure of depression symptoms over the past 2 weeks. Each of the 9 items is scored as 0 (not at all), 1 (several days), 2 (more than half the days) or 3 (nearly every day). Summing the 9 items the score range is 0-27. This instrument is validated in Spanish and will be used from two different approaches: as screening at baseline (PHQ-9 scoring <10: Negative test predictive value >95%) and to quantify depression severity over time (at 1, 6 and 12 months follow-up).
Anxious symptoms (GAD-7) | Base line, 1, 6 and 12 months follow-up
  Anxious symptoms will be measured by the GAD-7, which is also a reliable and valid 7-item measure of generalized anxiety symptoms, although it is also an effective screener for panic, social anxiety and posttraumatic stress disorders. Response options are similar to PHQ-9 (range from 0 = not at all, to 3 = nearly every day).Therefore, the total score ranges from 0-21. This instrument is validated in Spanish and will be used from two different approaches: as screening at baseline (GAD-7 scoring <10: Negative test predictive value >95%) and to quantify anxiety severity over time (at 1, 6 and 12 months follow-up).
Depression risk (predictD risk algorithm) | Baseline, 6 and 12 months follow-up
  The predictD risk algorithm (C-index = 0.82) assesses a series of risk factors for depression disorders, including: educational level, physical abuse in childhood, depression throughout life, number of serious problems in close people, and dissatisfaction with living at home. The predictD risk algorithm for Chile (C-index = 0.75) is very similar to the Spanish one, excluding three risk factors (dissatisfaction with unpaid work, physical abuse in childhood and number of serious problems in close people) and including a new one (satisfaction with the relationship with their partner). Both risk algorithms will be used to quantify the risk of depression overtime and will be assessed at baseline, at 6 and 12 months follow-up.
Anxiety risk (predictA risk algorithm) | Baseline, 6 and 12 months follow-up
  The predictA risk (C-index = 0.80) algorithm assesses the risk of anxiety in the next year. It includes a series of risk factors for anxiety disorders, including: sex, age, physical and mental quality of life, dissatisfaction with paid and unpaid work, financial difficulties, and medication for anxiety, depression or stress. This risk algorithm will be used to quantify the risk of anxiety overtime and will be assessed at baseline, at 6 and 12 months follow-up.
Physical and mental quality of life (SF-12) | Base line, 1, 6 and 12 months follow-up
  The SF-12 is included in both predictA and predictD risk algorithms and it is a valid a reliable instrument which gives measures of the physical and mental quality of life with a range of 0-100 points (higher score means better quality of life). The SF-12 will be assessed at baseline, and at 1, 6 and 12 months follow-up.
Acceptability and satisfaction with the Pandora app | 1 and 6 months follow-up
  Information on the use, adherence and acceptability of the Pandora intervention will be obtained automatically through the app. Some of these indicators are as follows: activity completion rates, completed assessments, amount of time spent in-app, frequency of use and number of log-ins.
  The U-MARS (User Version of the Mobile App Rating Scale) evaluates the quality and satisfaction of mobile health applications (Apps). The U-MARS consists of 27 items grouped into different domains: engagement, functionality, aesthetics, information quality and subjective quality. It uses a scale from 1 = "poor" to 5 = "excellent". Higher scores indicate better quality and satisfaction of the app. This measure will be assessed at 1 and 6 months follow-up.
Adverse effect (ad-hoc questionnaire) | 1 and 6 months follow-up
  An ad-hoc questionnaire will be designed to evaluate adverse effects arising from the Pandora app in order to gather information about any negative experiences or unintended consequences users may encounter while using the app. The primary purpose of this ad-hoc questionnaire is to capture user feedback on potential negative outcomes associated with the intervention (in general or due to a specific part of the intervention). Also, items of the questionnaire will assess how much that negative experience affects the wellbeing of the participants. This information will help in the future to make necessary adjustments to improve user experience, enhance safety features, and ensure that the app effectively supports users' health without causing harm. This measured will be assessed only at 1 and 6 months follow-up.

OTHER OUTCOMES:
Mediator: Physical activity (BPAQ-2) | Baseline, 1, 6 and 12 months follow-up
  Physical activity will be measured using the Brief Physical Activity Questionnaire (BPAQ-2), a widely used tool assessing adult physical activity levels. It includes two questions on frequency and duration of moderate- and vigorous-intensity activities over the past week. Based on responses, individuals are classified as low (insufficiently active), moderate (at least 150 minutes of moderate-intensity activity or equivalent), or high (at least 300 minutes of moderate-intensity activity or equivalent). Additionally, a subsample of 404 RCT participants (202 insufficiently active assigned to Pandora-1 and 202 assigned to usual care) will be assessed for physical activity over 7-day periods (24 hours per day) using Actigraph GT3X accelerometers at baseline, 1 and 6 months. Those participants classified as insufficiently active by the BPAQ-2 who were reclassified as active by accelerometers at baseline, will be excluded from this subsample of 404 participants of the PANDORA study.
Mediator: Insomnia (AIS-5) | Baseline, 1, 6 and 12 months follow-up
  Athens Insomnia Scale (AIS-5) aims to measure sleep induction, awakenings during the night, final awakening, total sleep duration and general sleep quality. Participants are asked to score each item from 0 (no problem at all) to 3 (very serious problem), if they have experienced any difficulty sleeping at least three times a week during the previous month (in order to fulfil the ICD-10 diagnostic criteria). Insomnia (AIS-5) will be assessed at baseline, 1, 6 and 12 months. A subsample of 404 RCT participants (202 sedentary individuals randomly assigned to Pandora-1 and 202 assigned to usual care) will be assessed for quantity and quality of sleep over 7-day periods (24 hours per day) using Actigraph GT3X accelerometers at baseline, 1 and 6 months.
Mediator: Social support (DUKE-UNC-11) | Baseline, 1, 6 and 12 months follow-up
  Social support will be measured by using an affective social support item and another confidential social support item from the DUKE- UNC-11 questionnaire, which were selected for having the highest item-subscale correlation coefficients in the Spanish validation of this questionnaire. A higher score on the social support-related items suggests that an individual feels more connected and supported by their social network, which is associated with better mental health outcomes. Conversely, lower scores may indicate feelings of loneliness or lack of support, which could be linked to higher levels of distress or poorer quality of life. This measure will be assessed at baseline, and at 1, 6 and 12 months follow-up.
Mediator: Perseverative thinking (PTQ-9) | Baseline, 1, 6 and 12 months follow-up
  Perseverative Thinking Questionnaire (PTQ) measures repetitive negative thinking (RNT) and has been translated (also in Spanish) and validated in several countries. RNT has been found to be involved in the development and maintenance of several types of emotional problems (including depression and anxiety disorders) and has therefore been suggested to be a transdiagnostic process. RNT was defined as a style of thinking about one's problem (current, past, or future) or negative experiences (past or anticipated) with three key characteristics: (1) being repetitive, intrusive, and uncontrollable; (2) perceived as unproductive; and (3) capturing mental resources. PTQ had good reliability (internal consistence and test-retest reliability) and validity (factorial and construct validity) and it was sensitive to change for the prevention of anxiety and depression. We will use the PTQ short version (9 items). The response to each item is given using a 5-point Likert scale from 0 = never to

CONTACTS AND LOCATIONS:
Locations (1):
- Juan Ángel Bellón Saameño, Málaga, Málaga, Spain